CLINICAL TRIAL: NCT03922204
Title: A Phase 1, Open-Label, Dose-Escalation, Safety, Tolerability, and Preliminary Efficacy Study of MCLA-145 in Participants With Advanced or Metastatic Malignancies
Brief Title: A Study of Bispecific Antibody MCLA-145 in Patients With Advanced or Metastatic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merus B.V. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCLA-145-CL01/MCLA-145-101; 2018-004396-13 (EudraCT Number)
Record Dates: First submitted 2019-04-15; First posted 2019-04-19 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Advanced Cancer; Solid Tumor, Adult; B-cell Lymphoma, Adult
Keywords: First-in-human; MCLA-145; Antibodies; Bispecific
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MCLA-145 (Experimental): In Part 1, the dose escalation phase, patients with advanced or recurrent/metastatic solid tumors or B-cell lymphomas will receive escalating doses of MCLA-145 (either Q2W for those patients in treatment at the time of Amendment #4 or Q3W with Amendment #4 approval). Treatment will be with MCLA-145 (monotherapy) for Group A, or in combination with pembrolizumab for Group B, until MTD or RDE is reached. In Part 2, the expansion phase, participants with advanced or metastatic solid tumors will receive intravenous infusion of MCLA-145 either in monotherapy (Group A) or in combination with pembrolizumab (Group B) at the recommended phase II dose every 3 weeks. The duration of each treatment cycle is 21 days
  Interventions: Drug: MCLA-145
- Group B Combination Treatment (Experimental): Patients in Group B will be treated with MCLA-145 in Combination with pembrolizumab 200mg Q3W.
  Interventions: Drug: MCLA-145; Drug: Pembrolizumab (Keytruda)

INTERVENTIONS:
Drug: MCLA-145 — full-length IgG1 bispecific antibody specifically targeting PD-L1 and CD137
  Other Names: bispecific
Drug: Pembrolizumab (Keytruda) — Group B patients will be treated in combination with MCLA-145 and pembrolizumab 200mg Q3W.
  Arms: Group B Combination Treatment

SUMMARY:
This is an open-label, non-randomized, Phase 1 study to determine the safety, tolerability, and preliminary efficacy of MCLA-145 in adult patients with advanced metastatic solid tumors or B-cell lymphomas. The study will be conducted in 2 parts.

DETAILED DESCRIPTION:
Study Design: This open label, multicenter, first in human study consists of 2 parts. Part 1 is a dose escalation to find the recommended dose of MCLA-145 in monotherapy or in combination with pembrolizumab.

Part 2 is a dose expansion to confirm the dose of MCLA-145, alone or in combination through further evaluation of safety, tolerability, Pk, preliminary antitumor activity, and functional target engagement.

The study includes three periods: Screening (up to 28 days prior to the first dose of study drug); Treatment (first dose of study drug with treatment cycles of 28 days for patients treated Q2W and 21 days for patients treated Q3W); Safety Follow-up (30 and 90 days after the last dose) including survival follow-up checks every 2 months up to 12 months after the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced or recurrent/metastatic solid tumors or B-cell lymphomas, that are considered non-amenable to surgery or other curative treatments or procedures (if applicable)
* Measureable disease per RECIST v1.1 or Lugano Criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Received prior standard therapy for advanced or recurrent/metastatic disease as applicable to tumor type
* Received a maximum of 4 prior systemic treatment regimens (inclusive of chemotherapy, immunotherapy, and targeted therapy regimens) for advanced or recurrent/metastatic disease
* Life expectancy of ≥12 weeks, as per investigator judgement

Exclusion Criteria:

* The following B-cell neoplasms: Burkitt lymphoma, lymphoblastic leukemia/lymphoma, lymphoplasmacytic lymphoma, chronic lymphocytic leukemia
* Prior therapy containing an anti-PD-L1 agent or T-cell agonist
* Current serious illness or medical condition including, but not limited to uncontrolled active infection
* Has not recovered to ≤ Grade 1 or baseline from toxic effects of prior therapy (including prior immunotherapy) and/or complications from prior surgical intervention before starting MCLA-145
* Prior ≥ Grade 3 immune-mediated AEs with anti-PD-1 therapy
* History of any grade immune-mediated ocular AEs.
* Known hypersensitivity or severe reaction to any component of MCLA-145 or formulation components
* Participants who have active or inactive autoimmune disease or syndrome (eg, rheumatoid arthritis, moderate or severe psoriasis, multiple sclerosis, inflammatory bowel disease) that has required systemic treatment in the past 2 years or who are receiving systemic therapy for an autoimmune or inflammatory disease (ie, with use of disease modifying agents, corticosteroids, or immunosuppressive drugs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with Dose Limiting Toxicities | first 28 days of treatment
Number of patients with Adverse Events and Serious Adverse Events | up to 90 days post-last dose

SECONDARY OUTCOMES:
Overall response rate (ORR) | Every 8 to 12 weeks until study ends, approximately 4 years
Duration of response ( DOR) | Every 8 to 12 weeks until study ends, approximately 4 years
Disease control rate ( DCR) | Every 8 to 12 weeks until study ends, approximately 4 years
Progression Free Survival ( PFS) | Every 8 to 12 weeks until study ends, approximately 4 years
Incidence of anti-drug antibodies against MCLA-145 | 12 months
Peak plasma concentration [Cmax] | 12 months
Area under the plasma concentration versus time curve [AUC] | 12 months
Half-life [t1/2] | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Laus, MD, Study Director — Merus B.V.
Locations (8):
- United States (3):
  - Moores Cancer Centre, La Jolla, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
- Belgium (2):
  - University Hospital Antwerp, Antwerp, Edegem
  - Universitair Ziekenhuis Gent, Ghent
- Netherlands Cancer Institute, Amsterdam, Netherlands
- Spain (2):
  - Hospital Universitario Fundarcion Jimenez Diaz, Madrid
  - Clinica Universidad de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: No